CLINICAL TRIAL: NCT00658697
Title: A Phase II Trial of Avastin, Docetaxel and Androgen Deprivation Followed by Continued Avastin and Androgen Deprivation for Men With a Rising Prostate Specific Antigen (PSA) After Local Therapy
Brief Title: Docetaxel, Bevacizumab and Androgen Deprivation Therapy After Definitive Local Therapy for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Mary-Ellen Taplin, MD, Associate Professor of Medicine, HMS, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-004
Record Dates: First submitted 2008-04-09; First posted 2008-04-15 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: Rising PSA; androgen deprivation; bevacizumab (avastin); docetaxel; lupron; zoladex; bicalutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Bevacizumab; Leuprolide; Goserelin; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel, Bevacizumab, and ADT (Experimental): Docetaxel:
  Intravenously given at 75 mg/m2 on day 1 of every 3 weeks for 4 cycles
  Bevacizumab:
  Intravenously given at (15 mg/kg) on day 1 of every 3 weeks for 8 cycles
  ADT or Luteinizing hormone-releasing hormone agonist (LHRH):
  Either subcutaneously or intramuscularly every three months for a total of 6 doses (total of 18 months)
  Bicalutamide:
  Oral Bicalutamide on day 84 once daily (after completing docetaxel, at 3 month) at dose of 50 mg for a total 15 months (4-18 months)
  Interventions: Drug: Docetaxel; Drug: Bevacizumab; Drug: ADT; Drug: Bicalutamide

INTERVENTIONS:
Drug: Docetaxel — Intravenously given at 75 mg/m2 on day 1 of every 3 weeks for 4 cycles
  Other Names: Taxotere, Docecad
Drug: Bevacizumab — Intravenously given at (15 mg/kg) on day 1 of every 3 weeks for 8 cycles
  Other Names: Avastin
Drug: ADT — Either subcutaneously or intramuscularly every three months for a total of 6 doses (total of 18 months)
  Other Names: Lupron or Zoladex
Drug: Bicalutamide — Starting on day 84 orally once daily until hormone therapy is completed
  Other Names: Casodex, Cosudex, Calutide, Kalumid

SUMMARY:
In this research study, we aim to evaluate the feasibility, toxicity and efficacy of early multimodality systemic therapy (a combination of docetaxe, bevacizumab, and androgen deprivation therapy(ADT) in men with biochemical recurrence (BCR) or who have a rising Prostate Specific Antigen (PSA) after treatment of their prostate cancer with surgery or radiation)

DETAILED DESCRIPTION:
A single arm phase 2 study designed to evaluate the rate of patients free from Prostate Specific Antigen (PSA) progression (TTP) one year after completing ADT for men with BCR after definitive local therapy for prostate cancer.

The null and alternative TTP rate were 41% and 60% respectively. A sample size of 42 would provide 80% power to detect the difference with a 2-sided type I error rate of 0.05.'

The primary objective was to evaluate the proportion of patients free from PSA progression after completing one year of ADT

The secondary objectives included

1. PSA response (< 0.2 ng/mL and < 0.01) at completion of docetaxel/bevacizumab, at completion of ADT and one year off ADT
2. Correlation of PSA response and TTP
3. Toxicity
4. Testosterone recovery at 6, 12 months off ADT

Treatment schedule details are as follows:

* Each treatment cycle lasts three weeks. During the first three months, participants will receive the Avastin and docetaxel on day 1 of each three-week cycle for a total of four doses of docetaxel/Avastin. Avastin and docetaxel are administered intravenously. The Avastin will continue to be given every three weeks after the docetaxel is completed for a total of 17 doses (one year) of Avastin therapy.
* Participants will receive zoladex (or lupron) on day 1 of the first cycle and then every 3 months for a total of 18 months. Zoladex is administered subcutaneously and Lupron is administered intramuscularly.
* Bicalutamide pills will be started at the completion of docetaxel chemotherapy (start of month 4) and will be taken once daily until hormone therapy is completed (total of 15 months).
* During all treatment cycles, the participant will have a physical exam and will be asked questions about their general health and specific questions about any problems they might be experiencing. Blood work will be performed every three weeks for the first three months and then every three months while on hormone therapy and during follow-up.
* After the final treatment participants will have a follow-up visit every three months for the first two years, every 4 months for the third year and every 6 months for years 4 and 5.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* History of biopsy documented prostate cancer (any Gleason score)
* Past treatment with prostatectomy with our without salvage prostate/pelvic radiation or primary radiation
* If past prostatectomy, pathologic stage no greater than T1-3, N1, M0
* PSA recurrence with PSAdt 8 months or less. There is no minimum PSA for prostatectomy patients. For patients treated with primary radiation therapy PSA should be 2.0ng/ml or greater
* No evidence of recurrent disease on exam, bone scan, CT/MRI abdomen/pelvis on CXR
* Prior ADT allowed if less than 6 months and testosterone recovered to within 50 units of normal range
* ECOG Performance status of 0-1
* Absolute neutrophil count of 1,500 mm3 or greater
* Platelet Count 100,000 mm3 or greater
* Total bilirubin within normal limits
* HG 8gm/dl or greater
* Testosterone within 50 units of normal range
* No history of bleeding or thromboses within the last 12 months that required medical intervention

Exclusion Criteria:

* History of cancer within 5 years, other than prostate cancer and non-melanoma skin cancer
* Medical condition requiring concomitant corticosteroids
* Active infection
* Prior chemotherapy
* Neuropathy requiring medical therapy
* Documented local recurrence or metastatic prostate cancer
* Inability to comply with study and/or follow-up procedures
* Life expectancy of less than 2 years
* Current, recent (within 4 weeks of first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored Avastin cancer study
* Inadequately controlled hypertension
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* NYHA Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 12 months prior to study enrollment
* History of stroke or transient ischemic attack at any time
* Known CNS disease
* Significant vascular disease
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening
* Known hypersensitivity to any component of Avastin

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-06; Primary Completion 2014-09 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - University of Maryland - Greenebaum Cancer Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 patients were enrolled between June 2, 2008 to December 14, 2010 at Dana Farber Cancer Institute and University of Michigan. One patient never started any study treatment, and was excluded from analysis.
Groups:
- Docetaxel, Bevacizumab, and ADT: Docetaxel:
  Intravenously given at 75 mg/m2 on day 1 of every 3 weeks for 4 cycles
  Bevacizumab:
  Intravenously given at (15 mg/kg) on day 1 of every 3 weeks for 8 cycles
  ADT or Luteinizing hormone-releasing hormone agonist (LHRH):
  Either subcutaneously or intramuscularly every three months for a total of 6 doses (total of 18 months)
  Bicalutamide:
  Oral Bicalutamide on day 84 once daily (after completing docetaxel, at 3 month) at dose of 50 mg for a total 15 months (4-18 months)
  Docetaxel
  Bevacizumab: intravenously given at (15 mg/kg) on day 1 of every 3 weeks for 8 cycles
  ADT: Either subcutaneously or intramuscularly every three months for a total of 6 doses (total of 18 months)
  Bicalutamide: Starting on day 84 orally once daily until hormone therapy is completed
Period: Overall Study
Arm/Group | Docetaxel, Bevacizumab, and ADT
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 41 (One patient never started any study treatment, and was excluded from analysis).
Groups:
- Docetaxel, Bevacizumab, and Androgen Deprivation Therapy (ADT): Docetaxel:
  Intravenously given at 75 mg/m2 on day 1 of every 3 weeks for 4 cycles
  Bevacizumab:
  Intravenously given at (15 mg/kg) on day 1 of every 3 weeks for 8 cycles
  Androgen deprivation therapy (ADT) or Luteinizing hormone-releasing hormone agonist (LHRH):
  Either subcutaneously or intramuscularly every three months for a total of 6 doses (total of 18 months)
  Bicalutamide:
  Oral Bicalutamide on day 84 once daily (after completing docetaxel, at 3 month) at dose of 50 mg for a total 15 months (4-18 months)
  Docetaxel
  Bevacizumab: intravenously given at (15 mg/kg) on day 1 of every 3 weeks for 8 cycles
  ADT: Either subcutaneously or intramuscularly every three months for a total of 6 doses (total of 18 months)
  Bicalutamide: Starting on day 84 orally once daily until hormone therapy is completed
Arm/Group | Docetaxel, Bevacizumab, and Androgen Deprivation Therapy (ADT)
Number analyzed (Participants) | 41
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [55 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Secondary Outcome: Proportion of Patients With PSA Responses at One Year After the Completion of ADT
Description: The PSA response was defined using two cut-offs: PSA <0.2 ng/mL or PSA <0.01 ng/mL at the one year after completion of ADT.
Time Frame: 1 year + 3 month off last ADT injection
Population: The analysis comprised of all patients received at least one treatment and had PSA data available* for the assessment of PSA responses at one year after completing ADT
  *Note excluded 5 patients started treatments but had no PSA information at one year.
Measure: Number (95% Confidence Interval); unit: percentage of participants with data
Groups:
- Docetaxel, Bevacizumab, and ADT: Docetaxel:
  Intravenously given at 75 mg/m2 on day 1 of every 3 weeks for 4 cycles
  Bevacizumab:
  Intravenously given at (15 mg/kg) on day 1 of every 3 weeks for 8 cycles
  ADT or Luteinizing hormone-releasing hormone agonist (LHRH):
  Either subcutaneously or intramuscularly every three months for a total of 6 doses (total of 18 months)
  Bicalutamide:
  Oral Bicalutamide on day 84 once daily (after completing docetaxel, at 3 month) at dose of 50 mg for a total 15 months (4-18 months)
  Docetaxel: Intravenously given at 75 mg/m2 on day 1 of every 3 weeks for 4 cycles
  Bevacizumab: Intravenously given at (15 mg/kg) on day 1 of every 3 weeks for 8 cycles
  ADT: Either subcutaneously or intramuscularly every three months for a total of 6 doses (total of 18 months)
  Bicalutamide: Starting on day 84 orally once daily until hormone therapy is completed
Arm/Group | Docetaxel, Bevacizumab, and ADT
Number analyzed (Participants) | 36
percentage of participants with data
  PSA <0.2 ng/mL | 44 [28 to 62]
  PSA <=0.01 ng/mL | 25 [12 to 42]

2. Secondary Outcome: Time to PSA Progression (TTP)
Description: For prostatectomy patients: at least two serial rising PSA from treatment nadir and PSA > 0.2 ng/mL. For patient receiving radiation therapy alone as primary local therapy, at least two serial rising PSA from treatment nadir and PSA > 2.0 ng/mL. Any new site of metastatic disease on imagining would be considered progression regardless of PSA value
Time Frame: participants were followed for the duration of the study, an average of 2 years
Population: the analysis dataset is comprised of all treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel, Bevacizumab, and ADT
Number analyzed (Participants) | 41
months | 27.5 [26 to 38]

3. Secondary Outcome: Testosterone Recovery
Description: Testosterone recovery was defined as >100 or within DFCI institute normal range (240-950) at one year after the completion of ADT
Time Frame: 2 years
Population: All treated patients with assessable testosterone level data
Measure: Number (95% Confidence Interval); unit: percentage of participants with data
Arm/Group | Docetaxel, Bevacizumab, and ADT
Number analyzed (Participants) | 35
percentage of participants with data
  Testosterone >=100 ng/mL | 83 [66 to 93]
  Testosterone >=240 ng/mL | 35 [31 to 66]

4. Primary Outcome: Prostate-Specific Antigen (PSA) Progression at 1 Year After Completing Androgen Deprivation Therapy (ADT)
Description: For prostatectomy patients: at least two serial rising PSA from treatment nadir and PSA > 0.2 ng/mL.
  For patient receiving radiation therapy alone as primary local therapy, at least two serial rising PSA from treatment nadir and PSA >2.0 ng/mL.
  Any new site of metastatic disease on imagining would be considered progression regardless of PSA value Clinical assessments (Vitals, Physical Exam, Performance Status, PSA and testosterone) were performed every 3 months starting at completion of hormone therapy until PSA progression.
Time Frame: participants were followed for the duration of the study, an average of 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants with data
Arm/Group | Docetaxel, Bevacizumab, and ADT
Number analyzed (Participants) | 41
percentage of participants with data | 98 [93 to 100]

5. Secondary Outcome: Toxicity
Description: Treatment related adverse events were graded based on CTCAE v. 3.0.
Time Frame: Assessed each cycle throughout treatment form time of first dose to 30 days post-treatment, up to 2 years
Population: All patients received at least one study therapies
Measure: Number; unit: participants
Groups:
- Docetaxel, Bevacizumab, and ADT: Docetaxel: Intravenously given at 75 mg/m2 on day 1 of every 3 weeks for 4 cycles
  Bevacizumab: Intravenously given at (15 mg/kg) on day 1 of every 3 weeks for 8 cycles
  ADT or Luteinizing hormone-releasing hormone agonist (LHRH): Either subcutaneously or intramuscularly every three months for a total of 6 doses (total of 18 months)
  Bicalutamide: Oral Bicalutamide on day 84 once daily (after completing docetaxel, at 3 month) at dose of 50 mg for a total 15 months (4-18 months)
  Docetaxel
  Bevacizumab: ntravenously given at (15 mg/kg) on day 1 of every 3 weeks for 8 cycles
  ADT: Either subcutaneously or intramuscularly every three months for a total of 6 doses (total of 18 months)
  Bicalutamide: Starting on day 84 orally once daily until hormone therapy is completed
Arm/Group | Docetaxel, Bevacizumab, and ADT
Number analyzed (Participants) | 41
participants
  Grade 3 treatment related AE | 16
  Grade 4 treatment related AEs | 5

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment form time of first dose and up to day 30 post-treatment, up to 2 years.
Arm/Group | Docetaxel, Bevacizumab, and ADT
Serious Adverse Events (participants affected / at risk) | 21/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel, Bevacizumab, and ADT (N=41)
Leukoencephalopathy (Nervous system disorders) | 1
Hematologic-other (Blood and lymphatic system disorders) | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Lower GI= hemorrhage NOS (Gastrointestinal disorders) | 1
Stomach= hemorrhage (Gastrointestinal disorders) | 1
Injection site reaction (General disorders) | 1
Allergic reaction (Immune system disorders) | 1
Perforation= appendix (Infections and infestations) | 1
Infection Gr0-2 neut= muscle (Infections and infestations) | 1
Infection Gr0-2 neut= wound (Infections and infestations) | 1
Leukocytes (Investigations) | 2
Neutrophils (Investigations) | 11
Hyponatremia (Metabolism and nutrition disorders) | 1
Neurologic-other (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel, Bevacizumab, and ADT (N=41)
Hemoglobin (Blood and lymphatic system disorders) | 1
Sinus arrhythmia (Cardiac disorders) | 1
Endocrine-other (Endocrine disorders) | 1
Vision-blurred (Eye disorders) | 1
Tearing (Eye disorders) | 9
Constipation (Gastrointestinal disorders) | 4
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 5
Hemorrhoids (Gastrointestinal disorders) | 1
Muco/stomatitis by exam= oral cavity (Gastrointestinal disorders) | 6
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 2
GI-other (Gastrointestinal disorders) | 1
Anus= hemorrhage (Gastrointestinal disorders) | 1
Oral cavity= hemorrhage (Gastrointestinal disorders) | 2
Rectum= hemorrhage (Gastrointestinal disorders) | 4
Abdomen= pain (Gastrointestinal disorders) | 2
Oral cavity= pain (Gastrointestinal disorders) | 3
Stomach= pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 35
Fever w/o neutropenia (General disorders) | 2
Rigors/chills (General disorders) | 1
Edema limb (General disorders) | 7
Edema trunk/genital (General disorders) | 1
Pain-other (General disorders) | 3
Flu-like syndrome (General disorders) | 2
Allergic reaction (Immune system disorders) | 8
Infection Gr0-2 neut= oral cavity (Infections and infestations) | 1
Infection Gr0-2 neut= skin (Infections and infestations) | 1
Infection w/ unk ANC dental-tooth (Infections and infestations) | 1
Infection w/ unk ANC upper airway NOS (Infections and infestations) | 1
Infection-other (Infections and infestations) | 1
Leukocytes (Investigations) | 4
Neutrophils (Investigations) | 2
Weight gain (Investigations) | 3
Weight loss (Investigations) | 1
Alkaline phosphatase (Investigations) | 1
ALT= SGPT (Investigations) | 5
AST= SGOT (Investigations) | 6
Creatinine (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1
Muscular/skeletal hypoplasia (Musculoskeletal and connective tissue disorders) | 1
Back= pain (Musculoskeletal and connective tissue disorders) | 1
Buttock= pain (Musculoskeletal and connective tissue disorders) | 2
Extremity-limb= pain (Musculoskeletal and connective tissue disorders) | 3
Joint= pain (Musculoskeletal and connective tissue disorders) | 6
Muscle= pain (Musculoskeletal and connective tissue disorders) | 4
Taste disturbance (Nervous system disorders) | 19
Mental status (Nervous system disorders) | 1
Neuropathy CN V jaw / face-sensory (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 12
Neurologic-other (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 12
Insomnia (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 4
Libido (Psychiatric disorders) | 4
Proteinuria (Renal and urinary disorders) | 3
Incontinence urinary (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1
Breast= pain (Reproductive system and breast disorders) | 1
Scrotum= pain (Reproductive system and breast disorders) | 1
Testicle= pain (Reproductive system and breast disorders) | 1
Erectile impotence (Reproductive system and breast disorders) | 4
Gynecomastia (Reproductive system and breast disorders) | 2
Sexual/Reproductive function-Other (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4
Nose= hemorrhage (Respiratory, thoracic and mediastinal disorders) | 17
Throat/pharynx/larynx= pain (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Nasal cavity/paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 19
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 11
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 1
Skin-other (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 16
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 31
Hematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes